CLINICAL TRIAL: NCT03053531
Title: Hearing Resources and Outcomes in the Emergency Department (HERO-ED)
Acronym: HERO-ED
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-01171
Record Dates: First submitted 2017-02-03; First posted 2017-02-15 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: Single-group study, with no control or comparison group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- HERO-ED RCT (Experimental): Subjects will be instructed on use of the HAD. The model that we will use is the PockeTalker Mini-Cog. This is a small (9.0cm X 5.5cm X 2.0cm) battery-powered electronic box that can be worn around the neck which connects via wires to both earphones and headphones (we will supply both earpieces, and let the patient choose). The RA, trained on use of the HAD by an experienced research audiologist, will instruct the patient in use of the HAD, and test the device to ensure proper functioning. The patient will also receive an instruction sheet (Appendix 3). Subjects will be encouraged to use the HAD during any encounters with ED staff.
  Interventions: Device: PockeTalker" Hearing Assistive Device (HAD)

INTERVENTIONS:
Device: PockeTalker" Hearing Assistive Device (HAD) — Investigators will test impacts of the provision of the HAD on hearing and understanding, and preparation for discharge. Just prior to going home, consented subjects will answer a set of survey questions, using an electronic tablet to support impaired hearing.

SUMMARY:
The Hearing Resources and Outcomes in the Emergency Department Pilot (HERO-ED Pilot), gathers preliminary data and hones procedures and measures, prior to undertaking HERO-ED. Since the HERO-ED Pilot does not involve random assignment (no control group), it will not test device effectiveness. However, the HERO-ED Pilot will test device acceptability and use. It will also provide preliminary data on, and allow us to fine-tune, the measures of effectiveness that we plan to use in HERO-ED

DETAILED DESCRIPTION:
The objectives are:

1. Measure the feasibility of in-ED hearing screening using HHIE-S and a handheld audiometer, among low-acuity11 ED patients age ≥75 years, by quantifying the proportion of eligible patients who complete hearing screening.
2. Test whether low-acuity older ED patients who screen positive for significant hearing loss (> 40 dB HL bilaterally and HHIE-S > 24) and are provided a hearing assistance device (HAD) use that device during the ED visit.
3. Test whether patients who are given a hearing assistance device will report ability as opposed to disability in hearing and understanding, using a six-item questionnaire adapted from a study by Cox et al.
4. Test whether those who are given a hearing assistance device will report being prepared for post-discharge care, using an adapted subset of the Care Transitions Measures (CTM).
5. Assess patient understanding of the HAD survey items within the post-use survey.

ELIGIBILITY:
Inclusion Criteria:

* low acuity clinical presentation (Emergency Severity Index11 triage criteria of 4 or 5, which indicates a high likelihood of being discharged home from the Emergency Department).
* Patients using hearing aids will not be excluded.

Exclusion Criteria:

* Lack of capacity to consent, as defined by the patient's ability to satisfactorily answer the questions outlined in the Evaluation to Sign Consent form (ESC) mentioned in the protocol. A legal representative/family member will not be able to consent for the patient in this study.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
Measure the feasibility of in-ED hearing screening using HHIE-S | 5 Minutes
  The HHIE-S is a ten-item survey and takes five minutes to complete. Responses to the HHIE reflect the extent to which hearing loss "feels" like a problem. Each response is scored on a 4, 2, or 0 point scale (4 = yes, 2 = sometimes, and 0 = no) for a maximum score of 40. A high score indicates high likelihood of hearing loss. Scores above 24 indicate a high likelihood of hearing loss and high adherence to HAD use

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Chodosh, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Medical Center, New York, New York, United States